CLINICAL TRIAL: NCT03669497
Title: Hypo-fractionated Radiotherapy Schedule of 26 GY in 5 Fractions With Simultaneous Integrated Boost (6 GY) in Advanced Incurable Breast Cancer: A Prospective Phase I/II Study (HYPORT-B).
Brief Title: Hypo-Fractionated Radiotherapy in Breast Cancer
Acronym: HYPORT-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/TMC/108/17
Record Dates: First submitted 2018-04-02; First posted 2018-09-13 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Palliative Radiotherapy; Hypo-fractionated Radiotherapy; Simultaneous integrated boost
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo fractionated radiotherapy (Experimental): Hypo fractionated whole breast radiotherapy with simultaneous integrated boost to the tumour
  Interventions: Radiation: Hypo fractionated whole breast radiotherapy

INTERVENTIONS:
Radiation: Hypo fractionated whole breast radiotherapy — Hypo fractionated radiotherapy to the whole breast and SCF to a dose of 26 GY in 5 fractions with simultaneous integrated boost in advanced incurable breast cancer

SUMMARY:
This is a prospective interventional phase I/II study which will be done at Tata Medical Centre, Kolkata. Total 30 eligible female patients, ≥18 years of age, with locally advance invasive carcinoma of breast, not amenable to curative surgery of metastatic breast cancer, planned for palliative loco regional radiotherapy will be enrolled in the study amongst which patients with left sided breast cancer (at least 10) will be recruited to study the feasibility of voluntary breath hold technique for heart sparing. Once consented, all patients will have regional baseline PET-CT scan of breast and tissue biopsy along with blood sampling done before studying radiotherapy. Planning Ct scan will then be taken, with standard planning CT scan for right breast cancers with implementation voluntary breath hold technique for the left breast disease. All patients will be treated with hypo-fractionated radiotherapy with schedule of 26Gy on 5 Fractions over 1 week with 6Gy simultaneously integrated boost with incorporation of breath hold technique for left breast disease. All patients will be assessed weekly during course of radiotherapy. The toxicity will be assessed using CTCAE version 4 and LENT SOMA toxicity criteria and the impact of the hypo-fractionated breast radiotherapy schedule on quality of life in advanced incurable breast cancer patients using FACT B scores PHQ4 questionnaire will also be assessed during treatment and follow-ups tissue bio0psy will be taken after 2 hours of completion of 1 st and last fraction of radiotherapy and biobanked for future radiobiological tests. Response evaluation will be done clinically and by regional PET CT scan using PERSIST criteria in 3 months after completion of radiotherapy. After completion of treatment, patient will initially be followed up every month for 1 st three months thereby 3 monthly for 2 years and 6 monthly for next 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * Female
  * Invasive carcinoma of the breast
  * ECOG performance status 0-2
  * Locally advanced breast cancer which is not amenable to curative surgery as decided by multidisciplinary tumour board.
  * Metastatic breast cancer patients:

    * Who are awaiting palliative locoregional radiotherapy for symptom (pain bleeding, ulceration, impending fungation) control.
    * Who have completed a scheduled course of palliative chemotherapy and is felt to benefit from local radiation therapy
  * Able to give informed consent

Exclusion Criteria:

* Breast reconstruction using implants

  * Concurrent cyto-toxic chemotherapy
  * Prior radiation to the chest wall / breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTCAE v 4.03) | 3 months
  Proportion of patients with Grade 3 or more toxicity at 3 months evaluated as per the CTCAE v 4.03 criteria.

SECONDARY OUTCOMES:
Response | 3 months
  To assess the response 3 months after radiotherapy clinically and by regional PET-CT scan using PERCIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjoy Chatterjee, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No